CLINICAL TRIAL: NCT05480228
Title: EPPIC-Net EN21-01 A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of 80 mg Daily of NRD135S.E1 Versus Placebo in Adult and Elderly Participants With Painful Diabetic Peripheral Neuropathy.
Brief Title: EPPIC-Net: Novaremed Painful Diabetic Peripheral Neuropathy ISA
Acronym: EN21-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James P. Rathmell, MD (Other)
Collaborators: New York University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, James P. Rathmell, MD, Chair, Department of Anesthesiology, Perioperative and Pain Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022P002381 (EN21-01); OT2NS122680-01 (NIH)
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: This study is an interventional, prospective, parallel-group, multicenter, randomized, double-blind, placebo-controlled, Phase 2 study.
Who Masked: Participant, Investigator
Masking Description: Randomization assignment will be blinded from study participants, staff from clinical sites, investigators, asset owner, IND sponsors, and/or designees.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NRD135S.E1 80mg/day (Experimental): NRD135S.E1 as a potential treatment for moderate to severe painful diabetic peripheral neuropathy (PDPN). While the activity of NRD135S.E1 has been extensively studied, its molecular target is not known, though it does not appear to work through any of the opioid receptors or molecular pathways currently targeted by available analgesics. The best evidence suggests it may act, at least in part, through modulating the Lyn kinase signaling pathway In clinical studies, NRD135S.E1 has been well tolerated at all dose levels tested in single-dose (up to 1,200 mg) and repeat-dose regimens (up to 300 mg/day over 5 days or 150 mg over 3 weeks), and it has been shown to have predictable pharmacokinetics with dose-dependent increases in exposure.
  Interventions: Drug: NRD135SE.1
- Matching placebo (Placebo Comparator): A matching placebo comparator will be used.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NRD135SE.1 — The double-blind treatment phase is up to 13 weeks.
  Other Names: NRD135s.E1, a small chemical entity for treatment of neuropathic pain
  Arms: NRD135S.E1 80mg/day
Other: Placebo — A matching placebo will be taken for up to 13 weeks.
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of the current hard gelatin capsule formulation of NRD135S.E1 80 mg once daily in the treatment of PDPN when administered for 13 weeks.

DETAILED DESCRIPTION:
This ISA describes a double-blind Phase II study of the PK/PD, safety, tolerability, and effect of 13 weeks of NRD135S.E1 (80mg/day) as an ISA within the context of the Platform Protocol to Assess Treatments for Painful Diabetic Peripheral Neuropathy, EN21-PP. The ISA is intended to be read and interpreted within the context of the Platform Protocol and focuses on the description of design features that are specific to NRD135S.E1.

ELIGIBILITY:
7.1 ISA-Specific Inclusion Criteria (To be used in conjunction with Platform Protocol criteria; note, some ISA criteria may be more stringent than Platform criteria; always follow the more stringent criteria when determining eligibility.)

1. Provides written consent for the EN21-01 ISA. Legally Authorized Representatives (LARs) are not allowed, but impartial witnesses may be utilized as needed for visually impaired participants.
2. Patient-reported daily 11-point NRS (for average pain over the last 24 hours) meets the criteria specified in "Appendix B: Blinded Information" during both the 7-day screening and 7-day baseline periods. The algorithm will be assessed centrally.

Waivers to the inclusion criteria will not be allowed. 7.2 ISA-Specific Exclusion Criteria (To be used in conjunction with Platform Protocol criteria; note, some ISA criteria may be more stringent than Platform criteria; always follow the more stringent criteria when determining eligibility.) Participants fulfilling any of the following criteria are not eligible for the study.

1. Diagnosis of alcohol or substance abuse or dependence (other than nicotine or caffeine) within the 2 years before the Screening visit. **This criterion is more stringent than a related Platform Protocol criterion.**
2. Moderate or severe renal impairment, known (documented) or defined as an estimated/calculated creatinine clearance/estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2, according to the Chronic Kidney Disease Epidemiology Collaboration formula during the screening process. **This criterion is more stringent than a related Platform Protocol criterion.**
3. Any of the following conditions related to corrected QT intervals using Fridericia's formula (QTcF):

   1. A QTcF > 500 ms prior to starting IP, up to and including the V3 pre-dose ECG.
   2. A history of the following additional risk factors for torsade de pointes: heart failure, hypokalemia, history or family history of long QT syndrome.
4. History of myocardial infarction, other clinically active significant heart disease, or stroke. **This criterion is more stringent than a related Platform Protocol criterion.**
5. Participants known to have participated in four or more studies for investigational pain drugs.
6. Participants known to be non-responders to more than three previous neuropathic pain medications at adequate doses over at least 4 weeks. Adequate doses (given as total daily doses) are defined as follows: 1,800 mg gabapentin; 300 mg pregabalin; opioid analgesics 60 mg oxycodone equivalent or 200 mg tramadol; 75 mg amitriptyline or equivalent tricyclic antidepressant; 60 mg duloxetine; 150 mg venlafaxine.
7. Known hypersensitivity or contraindication to any excipients of the study drug formulation.
8. Taking prohibited medications as described in Appendix A, "Prohibited Medications."
9. Major depressive episode within the 6 months before screening and/or a history of diagnosed recurrent major depressive disorder within two years. Any of the following conditions related to suicidality:

   1. Any suicidal ideation with intent, with or without a plan, at screening, i.e., answering "yes" to questions 4 or 5 on the Suicidal Ideation section of the Baseline/Screening version of the Columbia-Suicide Severity Rating Scale (C-SSRS);
   2. Answering "yes" on any item of the Suicidal Behavior Section (except for the "non-suicidal self-injurious behavior") of the C-SSRS if this behavior occurred in the past 2 years;
   3. A lifetime history of suicide attempt (V1).
10. Previous known or possible exposure to NRD135S.E1.

Waivers to the exclusion criteria will not be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
To demonstrate that NRD135S.E1 80 mg daily is superior to placebo in relieving neuropathic pain associated with PDPN, after 13 weeks' treatment. | 13 weeks
  Change from Baseline to Week 13 in the weekly mean of the daily 24-hour average pain measured by Numeric Rating Scale (NRS) (abbreviated herein as WAP for weekly average pain). The NRS is a 0-10 scale, with 0 indicating no pain, and 10 being the worst possible pain.
The frequency (i.e. number of participants) with treatment emergent adverse events (TEAEs) reported in the time period defined by first administration of IP until 7 days after the last dose of IP. | 13 weeks
  A treatment-emergent adverse event (TEAE) is any AE temporally associated with the use of study treatment whether or not considered by the investigator as related to study treatment.

SECONDARY OUTCOMES:
Occurrence of 30% reduction of WAP from Baseline to Week 13. | 13 weeks
  Weekly Average Pain is abbreviated as WAP.
Occurrence of 50% reduction of WAP from Baseline to Week 13. | 13 weeks
  Weekly Average Pain is abbreviated as WAP.

OTHER OUTCOMES:
To assess the effect of NRD135S.E1 in comparison to placebo with respect to Pain Catastrophizing Scale - Short Form 6 (PCS-SF6) | 13 weeks
  Catastrophizing is a pain-specific psychosocial construct comprising cognitive and emotional processes such as helplessness, pessimism, rumination about pain-related symptoms, and magnification of pain reports. The PCS-SF6 is a 6-item, self-report measure of catastrophic thinking associated with pain. Scores range from 0-24, with higher scores indicating more catastrophizing.
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the Pain, Enjoyment, and General activity scale (PEG). | 13 weeks
  The PEG is a three-item (each scored 0-10) multidimensional pain measure designed and validated for use in primary care and other ambulatory clinic patients, as a practical and useful tool to improve assessment and monitoring of chronic pain in primary care.
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the PROMIS Physical Functioning Short-Form 6b | 13 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Functioning short form is a 6-item scale that is widely used in pain research. It is a unidimensional scale that shows broad coverage of the physical function construct, good construct validity, and high levels of temporal stability. The PROMIS Physical Function Scale is expressed as a T-score, with a population mean of 50 and SD of 10. Higher scores represent better physical functioning; possible T scores in this distribution range from 21 to 59 (PROMIS, 2020).
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the Pain Health Questionnaire (PHQ-2). | 13 weeks
  The 2-item PHQ-2 is a brief depression screening tool that correlates strongly with PHQ-9 scores and shows good sensitivity for identifying individuals with depressive disorders in the general population in a variety of medical samples. Scores range from 0-6, with higher scores indicating more depressive symptomatology.
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the Generalized Anxiety Disorder - 2 item scale (GAD-2). | 13 weeks
  The GAD-2 is a 2-item screening tool that is widely used to screen for clinically significant anxiety symptoms and anxiety disorders in clinical settings. It shows good sensitivity and specificity as a screening tool for anxiety disorders. Scores range from 0-6, with higher scores indicating more anxiety symptomatology.
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the Tobacco, Alcohol, Prescription medication, and other Substance use Tool (TAPS-1). | 13 weeks
  The TAPS-1 is the screening component of the TAPS tool and consists of a single stem question with four items covering the frequency of past-12-month use of tobacco, alcohol, and illicit drugs, and non-medical use of prescription medications. Scores range from 0-4; higher scores indicate a higher likelihood of problematic substance use. The TAPS-1 shows good sensitivity and specificity for identifying substance use disorders.
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the PROMIS Sleep Disturbance - 6A. | 13 weeks
  The PROMIS Sleep Disturbance short form is a convenient 6-item scale that correlates strongly with the longer forms. The PROMIS Sleep Disturbance Scale is expressed as a T-score, with a population mean of 50 and standard deviation (SD) of 10. Possible T scores in this distribution range from 31.7 to 76.1 (PROMIS, 2021).
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the Sleep Duration Scale. | 13 weeks
  A single-item scale measuring the duration of actual sleep a participant has gotten, on average, over the past month. Numerical responses will be provided in hours and minutes.
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the Opioid Use Questionnaire (OUQ). | 13 weeks
  The OUQ is an indicator of past or present use of any of the listed opioid medications. There are a total of three yes/no items where a yes indicates the use of such medications.
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the Patient Global Impression of Change (PGIC). | 13 weeks
  The PGIC is a single-item measure of patient-reported improvement that is widely used as a general outcome measure in studies of chronic pain patients. It is often used as an index of treatment-associated change, and patient-reported improvements in the form of PGIC scores correlate robustly with significant improvement in pain intensity, pain interference with activities of daily living, mood, and quality of life (Perrot and Lanteri-Minet, 2019).
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the Norfolk Quality of Life - Diabetic Neuropathy (Norfolk QOL-DN) | 13 weeks
  The Norfolk QOL-DN is a validated 47-item, patient-reported outcome measure, sensitive to the different features of diabetic neuropathy (DN) including small fiber, large fiber, and autonomic function. A higher score indicates higher levels of neuropathic pain.
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the Neuropathy examination. | 13 weeks
  The neuropathy examination will be a single procedure consisting of visual inspection of the feet, brief distal motor exam, ankle and knee deep tendon reflexes, and a standardized sensory exam. This exam will collect the data needed to calculate several common scores including: the Michigan Neuropathy Screening Instrument (MNSI) Part B, the Utah Early Neuropathy Scale (UENS) and the Toronto Clinical Scoring System (TCNS). The MSNI Part B consists of visual inspection of the feet and assessment of ankle reflexes, vibration sense, and monofilament testing. The TCNS is quantitative scoring system for evaluating the severity of peripheral neuropathy. Most of the test is done on or near the toes, light touch testing is done with a 10gm monofilament fiber. The UENS consists of testing the distal lower extremities for motor function, sharp sensation, allodynia, vibration sensation, and deep tendon reflexes. It is scored on a scale of 0-42 where zero is normal.
To assess the effect of NRD135S.E1 in comparison to placebo with respect to the actigraphy step count. | 13 weeks
  Mean daily step counts will be used as an index of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Robinson-Papp, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (26):
- United States (26):
  - University of California, San Diego, San Diego, California
  - South Lake Pain Institute, Clermont, Florida
  - SIMEDHealth LLC, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Northwestern Department of Neurology, Chicago, Illinois
  - Healthcare Research Network (Flossmoor), Flossmoor, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland - Baltimore, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - MGH Department of Anesthesia, Critical Care, and Pain, Boston, Massachusetts
  - Healthcare Research Network (Hazelwood), Hazelwood, Missouri
  - NYU Langone Manhattan, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center/Neurological Institute, New York, New York
  - University of Rochester, Rochester, New York
  - Clinical Inquest Center, Beavercreek, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Low Country Pain Center, Orangeburg, South Carolina
  - American Indian Clinical Trials Research Network, Rapid City, South Dakota
  - Nerve and Muscle Center of Texas, Houston, Texas
  - Clinicore International, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - VCU Department of Neurology, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No The use of Global Unique Identifiers (GUIDs) allows data to be linked with a given research participant, without revealing any of the participant's identifiable information. All participants in NIH-funded research must have a GUID. This study is using the Biomedical Research Informatics Computing System (BRICS) GUID platform to assign GUIDs. This ID should be generated at the time of Informed Consent since it requires several pieces of patient information (e.g., last name at birth, first name at birth, sex at birth, day, month and year of birth, city and country of birth, etc.). The GUID will be a combination of letters and numbers to form a unique identifier, e.g. TBIAC412JJK. Sites should maintain a list to link the GUID to the participant.

REFERENCES:
- [Background] Dworkin RH, Turk DC, Peirce-Sandner S, McDermott MP, Farrar JT, Hertz S, Katz NP, Raja SN, Rappaport BA. Placebo and treatment group responses in postherpetic neuralgia vs. painful diabetic peripheral neuropathy clinical trials in the REPORT database. Pain. 2010 Jul;150(1):12-16. doi: 10.1016/j.pain.2010.02.002. Epub 2010 Mar 3. No abstract available. PMID 20202753
- [Background] Tarpey T, Petkova E, Ciarleglio A, Ogden RT. Extracting scalar measures from functional data with applications to placebo response. Stat Interface. 2021;14(3):255-265. doi: 10.4310/20-sii633. PMID 34316322
- [Background] Tarpey T, Petkova E, Lu Y, Govindarajulu U. Optimal Partitioning for Linear Mixed Effects Models: Applications to Identifying Placebo Responders. J Am Stat Assoc. 2010 Jan 1;105(491):968-977. doi: 10.1198/jasa.2010.ap08713. PMID 21494314
- [Background] Van Buuren, S., & Groothuis-Oudshoorn, K. (2011). Journal of Statistical Software mice: Multivariate Imputation by Chained Equations in R (Vol. 45). http://www.jstatsoft.org/